CLINICAL TRIAL: NCT01535586
Title: A Randomized Cross Over Trial of Two Treatments for Obstructive Sleep Apnea in Veterans With Post Traumatic Stress Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The VA Western New York Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mr. Shawn Gall, Administrative officer, The VA Western New York Healthcare System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSR&D I01CX000478
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP; MAD; sleep apnea; PTSD
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Active Comparator): participants will be treated with continuous positive airway pressure (CPAP) for 12 weeks
  Interventions: Device: CPAP versus MAD
- MAD (Active Comparator): Participants will be treated with a mandibular advancing device for 12 weeks
  Interventions: Device: CPAP versus MAD

INTERVENTIONS:
Device: CPAP versus MAD — Cross over design

SUMMARY:
Sleep disturbances are cardinal features of Veterans with post traumatic stress disorder (PTSD). In particular, obstructive sleep apnea is reported to occur more frequently in patients with PTSD compared to those without PTSD and contribute to worsening cognitive and behavioral functions. Continuous positive airway pressure (CPAP) is considered the treatment of choice for OSA but adherence to CPAP in Veterans with PTSD is poor compared to the general population. The proposed study aims at comparing the efficacy, tolerability, and adherence of mandibular advancing devices-an alternative therapy to OSA- to CPAP. The study is instrumental in identifying the optimal OSA therapy for Veterans with PTSD and the OSA phenotype that would predict MAD response.

ELIGIBILITY:
Inclusion Criteria:

* • Consecutive patients aged 18-70 years of age

  * Documented obstructive sleep apnea by polysomnography (AHI≥5 or more/hr)
  * Established diagnosis of PTSD related to any past lifetime traumatic event and have a diagnosis of current, chronic PTSD

Exclusion Criteria:

* • Central sleep apnea defined as central apnea/hypopnea >50% of the total respiratory events

  * Prior treatment for sleep apnea
  * Veterans with fewer than 4 teeth remaining in either arch
  * Coexisting narcolepsy
  * Tempo-mandibular joint disease
  * Epilepsy
  * Prominent suicidal or homicidal ideation
  * Diagnosis of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 12 weeks
  The primary objective of this trial is to assess the efficacy of MAD versus CPAP in the treatment of OSA in Veterans with PTSD.Treatment will be considered efficacious (successful) when the apnea-hypopnea index is < 5 in the absence of hypoxemia defined as SvO2<90%.

SECONDARY OUTCOMES:
Adherence | 12 weeks
  Adequate adherence will be defined as device usage of >4 hr per night for 70% of days